CLINICAL TRIAL: NCT01394497
Title: Infusione Sistemica e Loco-regionale di N-Acetilcisteina Nel Prelievo di Fegato: Uno Studio Prospettico Randomizzato Controllato. Fase II.
Brief Title: Use of N-Acetylcysteine During Liver Procurement
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Azienda Ospedaliera di Padova (Other)
Responsible Party: Principal Investigator, Prof. Umberto Cillo, Director of the Hepatobiliary Surgery and Liver Transplantation Unit, Azienda Ospedaliera di Padova
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1635P
Record Dates: First submitted 2011-07-12; First posted 2011-07-14 (Estimated); Last update posted 2013-02-18 (Estimated); Status verified 2013-02

CONDITIONS: Liver Failure; Liver Failure, Acute; Liver Diseases; Carcinoma, Hepatocellular; Liver Neoplasms
Keywords: Liver Transplantation; Graft Survival; Graft Rejection; Primary Graft Dysfunction; Tissue and Organ Harvesting; Tissue and Organ Procurement; Tissue Donors; Cold Ischemia
MeSH Terms: conditions — Liver Failure; Liver Failure, Acute; Liver Diseases; Carcinoma, Hepatocellular; Liver Neoplasms; Primary Graft Dysfunction | interventions — Acetylcysteine; N-monoacetylcystine; halofantrine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NAC procurement protocol (Experimental): The allocated organ, in addition to the standard procedure, was treated with a systemic NAC infusion before initiating the liver harvesting procedure, and a loco-regional infusion into the portal vein before cross-clamping.
  Interventions: Drug: N-acetylcystein
- Standard procurement procedure (No Intervention): Allocated organ was treated according to the centre's standard procurement procedure: a modified double perfusion technique, where donor livers are gravity-perfused in situ via the aorta and portal vein with Celsior solution at 4 °C. After hepatectomy, donor livers were further perfused at the back-table with Celsior solution and then stored in conventional bags containing the same solution at 4 °C until transplantation.

INTERVENTIONS:
Drug: N-acetylcystein — 15 min systemic NAC infusion of the donor (30 mg/kg, maximum dose 3000 mg) diluted into 500 ml 5 % glucose solution, 30 min before initiating the liver harvesting procedure, and a loco-regional infusion (150 mg/kg of estimated liver weight, maximum dose 300 mg) into the portal vein 5 min before cross-clamping.
  Other Names: Fluimucil (Zambon, Italy); ACC (Hexal AG); Acemuc (Betapharm, Germany); Acetyst (Ristert, Germany); Acetadote (Cumberland Pharmaceuticals); Asist (Bilim Pharmaceuticals, Turkey); Brunac eyedrops (Bruschettini, Italy); Fluimukan (Lek, Slovenia); Flumil (Pharmazam, Spain); Lysox (Menarini); Mucinac (Cipla, India); Mucohelp (Neiss Labs, India); Mucolysin (Sandoz); Mucomelt (Venus Remedies, India); MUCOMIX (Samarth Life Sciences, India); Mucomyst (Bristol-Myers Squibb); Nytex (Pharos,Indonesia); Parvolex (GSK); PharmaNAC (BioAdvantex Pharma Inc., North America); Rheunac (Tree Of Life, Israel); Solmucaïne (IBSA, Switzerland); Trebon N (Uni-pharma)
  Arms: NAC procurement protocol

SUMMARY:
Randomized prospective study on the impact on the post-LT outcome by the infusion of N-acetylcysteine (NAC) during the liver procurement procedure, as an anti-oxidant agent to reduce the ischemia-reperfusion damage of organs for liver transplantation (LT).

DETAILED DESCRIPTION:
Anti-oxidant agents have the potential to reduce the ischemia-reperfusion damage of organs for liver transplantation (LT). In this randomized prospective study, we seek to study the impact on the post-LT outcome of the infusion of N-acetylcysteine (NAC) during the liver procurement procedure.

Potential grafts, assigned to adult candidates with chronic liver disease enlisted for first LT, will randomly be included in a one-to-one ratio with a sequential closed envelope single-blinded assignation procedure to either the NAC protocol or in the standard procedure (without NAC).

The NAC protocol comprises: a systemic NAC infusion (30 mg/kg) one hour before the beginning of liver procurement; a loco-regional NAC infusion (300 mg through the portal vein) just before cross-clamping.

ELIGIBILITY:
Inclusion Criteria:

* all consecutive subjects with chronic liver disease undergoing first Liver Transplantation receiving deceased donor livers

Exclusion Criteria:

* recipients with acute liver disease;
* paediatric patients or adult patients receiving a liver from a paediatric donor;
* patients undergoing multiple-organ transplantation;
* patients undergoing re-transplantation of the Liver;
* patients undergoing living donor Liver Transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2006-12; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Graft survival | up to 60 months

SECONDARY OUTCOMES:
Patient survival | up to 60 months
Primary graft dysfunction | up to 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Umberto Cillo, MD, Study Director — Azienda Ospedaliera di Padova; Francesco D'Amico, MD, Principal Investigator — Azienda Ospedaliera di Padova
Locations (1):
- Azienda Ospedaliera di Padova, Padua, Padova, Italy

REFERENCES:
- [Result] D'Amico F, Vitale A, Gringeri E, Valmasoni M, Carraro A, Brolese A, Zanus G, Neri D, Boccagni P, Violi P, Pauletto A, D'Amico FE, D'Amico DF, Cillo U. SYSTEMIC AND LOCO-REGIONAL INFUSION OF N-ACETILCISTEINA DURING LIVER PROCUREMENT: A PROSPECTIVE RANDOMIZED CONTROLLED STUDY (Abstract# 488), The International Liver Transplantation Society: 14th Annual International Congress, July 9-12, 2008, Paris, France. Liver Transplantation, 14: S1-S269. doi: 10.1002/lt.21569
- [Result] D'Amico F, Vitale A, Piovan D, Bertacco A, Ramirez Morales R, Chiara Frigo A, Bassi D, Bonsignore P, Gringeri E, Valmasoni M, Garbo G, Lodo E, D'Amico FE, Scopelliti M, Carraro A, Gambato M, Brolese A, Zanus G, Neri D, Cillo U. Use of N-acetylcysteine during liver procurement: a prospective randomized controlled study. Liver Transpl. 2013 Feb;19(2):135-44. doi: 10.1002/lt.23527. Epub 2012 Sep 26. PMID 22859317
- See also: Hepatobiliary surgery and Liver Transplantation Unit, University Hospital of Padua (Italy) — http://www.fegatochirurgia.com/